CLINICAL TRIAL: NCT07278193
Title: Combined Effects of Foam Rolling and Dynamic Stretching in Patients With Piriformis Syndrome
Brief Title: Foam Rolling and Dynamic Stretching in Piriformis Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Rabia Kanwal, PT, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOL/IREB/25/09/0047
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Piriformis Syndrome
Keywords: foam rolling; dynamic stretching; piriformis muscle; Quality of life
MeSH Terms: conditions — Piriformis Muscle Syndrome | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Model Description
Who Masked: Outcomes Assessor
Masking Description: Masking Description
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Foam Rolling): (Experimental): Participants will use a foam roller to apply pressure to the piriformis muscle and surrounding areas, targeting tight spots and trigger points. This technique helps release muscle tension, improve blood circulation, and alleviate pain by using slow, controlled rolling motions that will last 5-10 minutes twice daily, 3 sessions per week for up to 8 weeks.
  Interventions: Other: Group A (Foam Rolling)
- Group B (Foam rolling and Dynamic Stretching) (Experimental): Group B (Foam rolling and Dynamic Stretching): Group B will receive foam rolling with dynamic stretching. Hot pack will be applied 5-3 min before rolling and dynamic stretching. The rolling helps release muscle tension, improve blood circulation, and alleviate pain by using slow, controlled rolling motions will last 5-10 minutes. The stretching routine will include exercises like hip swings, seated piriformis stretches, and Dynamic Figure-Four Stretch supine stretch. Each stretching session will last 10-15 minutes and will be conducted twice daily (3 days a week) for 8 weeks. This approach ensures gradual improvement in muscle flexibility and joint mobility while maintaining participant safety and comfort throughout the intervention. Ultrasound therapy will be applied after stretching.
  Interventions: Other: Group B (Foam rolling and Dynamic Stretching)

INTERVENTIONS:
Other: Group A (Foam Rolling) — Foam Rolling Alone (FR) (~10 minutes)
  * Piriformis Foam Rolling: 30-60 sec per side (2-3 sets)
  * Glutes & Lower Back Foam Rolling: 30 sec each (2-3 sets)
  * Hamstrings & IT Band Foam Rolling: 30 sec each (2-3 sets) Focus: Slow, controlled rolling with sustained pressure on tender spots.
  Arms: Group A (Foam Rolling):
Other: Group B (Foam rolling and Dynamic Stretching) — Dynamic Stretching (~5-6 minutes)
  * Dynamic Piriformis Stretch: Standing knee-to-opposite-shoulder pull (10 reps per leg)
  * Leg Swings: Forward and sideways (10 reps each leg)
  * Walking Lunges with Rotation: 10 reps per leg
  * Hip Circles & Controlled Butt Kicks: 10 reps each
    3. Cool-Down (2-3 minutes) Objective: Reduce muscle tension and promote recovery.
  * Seated Piriformis Stretch: 30 sec hold per side (2 sets)
  * Hamstring Stretch: 30 sec hold per leg
  * Lower Back Stretch (Child's Pose): 30 sec
  Arms: Group B (Foam rolling and Dynamic Stretching)

SUMMARY:
To compare the combined effects of foam rolling and dynamic stretching in patients with piriformis syndrome.

1. Warm-Up (2-3 minutes) Objective: Increase blood flow and prepare muscles for stretching.

   * Marching in Place - 30 seconds
   * Pelvic Tilts - 10 reps
   * Gentle Hip Circles - 10 reps each direction
2. Intervention Phase (8-10 minutes) Group 1: Foam Rolling Alone (FR) (~10 minutes)

   * Piriformis Foam Rolling: 30-60 sec per side (2-3 sets)
   * Glutes & Lower Back Foam Rolling: 30 sec each (2-3 sets)
   * Hamstrings & IT Band Foam Rolling: 30 sec each (2-3 sets)

   Focus: Slow, controlled rolling with sustained pressure on tender spots. Group 2: Foam Rolling + Dynamic Stretching (FR+DS) (~10-12 minutes) Step 1: Foam Rolling (~5-6 minutes, same as Group 1) Step 2: Dynamic Stretching (~5-6 minutes)
   * Dynamic Piriformis Stretch: Standing knee-to-opposite-shoulder pull (10 reps per leg)
   * Leg Swings: Forward and sideways (10 reps each leg)
   * Walking Lunges with Rotation: 10 reps per leg
   * Hip Circles & Controlled Butt Kicks: 10 reps each
3. Cool-Down (2-3 minutes) Objective: Reduce muscle tension and promote recovery.

   * Seated Piriformis Stretch: 30 sec hold per side (2 sets)
   * Hamstring Stretch: 30 sec hold per leg
   * Lower Back Stretch (Child's Pose): 30 sec

Progression & Adjustments

* Gradual increase in duration or intensity as tolerated.
* Modify exercises if discomfort or pain occurs.
* After week 4, increase dynamic stretch duration if flexibility improves.

Outcome Measures

The effectiveness of the intervention will be assessed through the following key outcome measures:

1. Pain Level - Evaluating changes in discomfort intensity during daily activities and movement.
2. Range of Motion (ROM) - Measuring improvements in hip flexibility and mobility.

DETAILED DESCRIPTION:
To compare the combined effects of foam rolling and dynamic stretching in patients with piriformis syndrome.

Inclusion Criteria:

* Age 35-50 years diagnosed with Piriformis Syndrome based on clinical findings. (Chang et al., 2024)
* Having positive FAIR test is commonly used to diagnose piriformis syndrome.
* Pain intensity of at least 4 on the numeric pain rating scale (NPRS) at baseline(A Penichet-Tomas et al., 2021).

DIAGNOSTIC CRITERIA OF PIRIFORMIS SYNDROME

The diagnostic criteria for piriformis syndrome include clinical history, physical examination findings. The symptoms include buttock pain radiating to the posterior thigh or leg, worsened by sitting, climbing stairs, or activities that stretch the piriformis muscle. Physical examination, tenderness over the piriformis muscle or sciatic notch and a positive FAIR test (Flexion, Adduction, and Internal Rotation) are indicative. Additional tests, such as the Pace test and Straight Leg Raise with external rotation.

Exclusion Criteria:

* Current use of medications such as strong analgesics or muscle relaxants. (e.g., injections, surgery) within the last three months.
* Uncontrolled medical conditions, such as active infections, cancer, or cardiovascular issues that may interfere with the study or the participant's ability to complete the protocol safely(Alfonso Penichet-Tomas et al., 2021).
* History of lumbar disc herniation, spinal stenosis, or other serious lumbar spine pathologies that may cause similar symptoms.
* Prior surgeries in the lumbar spine, hip, or pelvis that may interfere with the study's outcomes(Pişirici et al., 2020).
* ASSESMENT TOOL
* Pain (NPRS): Pain will be measured using the NPRS (Numeric pain rating scale) which assesses the intensity of pain on a scale ranging from 0 no pain to 10 worst imaginable pain. Participants will report their pain levels at baseline and post-intervention to determine the efficacy of foam rolling and dynamic stretching.
* ROM (Goniometer):The piriformis muscle plays a crucial role in hip movement and stabilization. Its primary function is external rotation of the hip with a normal range of motion (ROM) of 0°-45°. Additionally, the piriformis assists in hip abduction with a typical range of 0°-45°. Interestingly, the piriformis also supports internal rotation with a normal ROM of 0°-35°. These movements are assessed using a goniometer to measure hip rotation, where improvements in internal and external rotation, as well as abduction ROM, indicate reduced piriformis tightness and enhanced hip flexibility
* SF-12 (QoL): The SF-12 (Short Form Health Survey) is a validated tool used to assess quality of life (QoL) across physical and mental health domains. It provides a concise yet comprehensive evaluation of functional limitations, pain, and overall well-being. Among individuals with piriformis syndrome, SF-12 can effectively measure the impact of pain and muscle tightness on daily activities and mental health.

Randomization: Randomization will be performed using a computer-generated method, ensuring that participants are randomly assigned to both groups. This process will minimize bias, and then half of the data will be allocated to each group for analysis.

Treatment Plan

Group A (Foam Rolling): Participants will use a foam roller to apply pressure to the piriformis muscle and surrounding areas, targeting tight spots and trigger points. This technique helps release muscle tension, improve blood circulation, and alleviate pain by using slow, controlled rolling motions that will last 5-10 minutes twice daily, 3 sessions per week for up to 8 weeks.

Group B (Foam rolling and Dynamic Stretching): Group B will receive foam rolling with dynamic stretching. Hot pack will be applied 5-3 min before rolling and dynamic stretching. The rolling helps release muscle tension, improve blood circulation, and alleviate pain by using slow, controlled rolling motions will last 5-10 minutes. The stretching routine will include exercises like hip swings, seated piriformis stretches, and Dynamic Figure-Four Stretch supine stretch. Each stretching session will last 10-15 minutes and will be conducted twice daily (3 days a week) for 8 weeks. This approach ensures gradual improvement in muscle flexibility and joint mobility while maintaining participant safety and comfort throughout the intervention. Ultrasound therapy will be applied after stretching.

Routine Physical Therapy

Duration: 8 weeks Frequency: Twice daily, 3 days a week Session Duration: 10-15 minutes per session

ELIGIBILITY:
Inclusion Criteria:

* Age 35-50 years diagnosed with Piriformis Syndrome based on clinical findings. (Chang et al., 2024)
* Having positive FAIR test is commonly used to diagnose piriformis syndrome.
* Pain intensity of at least 4 on the numeric pain rating scale (NPRS) at baseline(A Penichet-Tomas et al., 2021).

DIAGNOSTIC CRITERIA OF PIRIFORMIS SYNDROME

The diagnostic criteria for piriformis syndrome include clinical history, physical examination findings. The symptoms include buttock pain radiating to the posterior thigh or leg, worsened by sitting, climbing stairs, or activities that stretch the piriformis muscle. Physical examination, tenderness over the piriformis muscle or sciatic notch and a positive FAIR test (Flexion, Adduction, and Internal Rotation) are indicative. Additional tests, such as the Pace test and Straight Leg Raise with external rotation.

Exclusion Criteria:

* Current use of medications such as strong analgesics or muscle relaxants. (e.g., injections, surgery) within the last three months.
* Uncontrolled medical conditions, such as active infections, cancer, or cardiovascular issues that may interfere with the study or the participant's ability to complete the protocol safely(Alfonso Penichet-Tomas et al., 2021).
* History of lumbar disc herniation, spinal stenosis, or other serious lumbar spine pathologies that may cause similar symptoms.
* Prior surgeries in the lumbar spine, hip, or pelvis that may interfere with the study's outcomes(Pişirici et al., 2020).

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-01-02 (Estimated)

PRIMARY OUTCOMES:
Goniometer | At baseline, 4th week and 8th week
  Range of motion will be measured using the Goniometer. Its primary function is external rotation of the hip with a normal range of motion (ROM) of 0°- 45°additionally, the piriformis assists in hip abduction with a typical range of 0°-45°. Interestingly, the piriformis also supports internal rotation with a normal ROM of 0°-35°.
NPRS (Numeric pain rating scale) | Each outcome variable will be measured at baseline, mid-intervention and post-intervention
  Pain will be measured using the NPRS (Numeric pain rating scale) which assesses the intensity of pain on a scale ranging from 0 no pain to 10 worst imaginable pain. Participants will report their pain levels at baseline and post-intervention to determine the efficacy of foam rolling and dynamic stretching

SECONDARY OUTCOMES:
SF-12 (Short Form Health Survey) | At baseline, 4th week and 8th week
  The SF-12 (Short Form Health Survey) is a validated tool used to assess quality of life (QoL) across physical and mental health domains. It provides a concise yet comprehensive evaluation of functional limitations, pain, and overall well-being. Among individuals with piriformis syndrome, SF-12 can effectively measure the impact of pain and muscle tightness on daily activities and mental health (Zhou et al., 2024).

CONTACTS AND LOCATIONS:
Overall Officials: Sana Akram, MS-OMPT, Study Chair — University of Lahore
Locations (1):
- University of Lahore teaching hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No